CLINICAL TRIAL: NCT04878835
Title: Effects of Ranibizumab on Microvasculature, Oxidative Stress and Recurrence in Primary Pterygium Surgery
Brief Title: Effects of Ranibizumab in Primary Pterygium Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Kueh Yee Cheng, PhD, https://medic.usm.my/expertsppsp/kueh-yee-cheng, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USM/JEPeM/18010009
Record Dates: First submitted 2021-04-26; First posted 2021-05-10 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Patients With Primary Nasal Pterygium

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): No intervention was given. No intralesional ranibizumab (Lucentis; Genentech, Inc, San Francisco, California, USA 0.5mg/ 0.05mL) was given at 2 weeks prior to pterygium excision surgery
- Intervention group (Experimental): The interventional group was given intralesional ranibizumab (Lucentis; Genentech, Inc, San Francisco, California, USA 0.5mg/ 0.05mL) 2 weeks prior to pterygium excision surgery
  Interventions: Biological: intralesional ranibizumab

INTERVENTIONS:
Biological: intralesional ranibizumab — Lucentis; Genentech, Inc, San Francisco, California, USA 0.5mg/ 0.05mL
  Arms: Intervention group

SUMMARY:
Pterygium is a common ocular surface disease in Malaysia. Without treatment, it can lead to severe visual impairment. Recurrence is the commonest complication and novel treatment approaches are crucial to prevent vision loss. The biological processes underlying the formation of pterygium are complex, but central to its pathogenesis is the angiogenic cytokine vascular endothelial growth factor (VEGF). VEGF is upregulated under conditions of increased oxidative stress, which plays an integral role in pterygium development (Cardenas-Cantu et al., 2016, Karaman, 2018, Norrby, 1998, Rossino et al., 2020, Shibunya, 2011).Various biomarkers on pterygium have been identified and are useful to determine the effectiveness of new modality treatment for pterygium. These markers can be identified via histopathological stain such as Masson Trichrome to observe changes of collagen fibres. Other identifiable markers include the use of special immunohistochemical stain such as anti CD34 antibody for microvascular density and anti-8-OHdG antibody for oxidative changes in the pterygium tissue. By analyzing the changes with or without Ranibizumab injection in addition to observation of clinical recurrence rate of pterygium, we are able to conclude the effectiveness of anti-VEGF on pterygium recurrence. The aim of the study was to evaluate the association between collagen fibres changes, microvascular density changes and inflammation resultant from oxidative stress with the clinical recurrence of pterygium following intralesional Ranibizumab injection in comparison to control group.

DETAILED DESCRIPTION:
This is a prospective interventional study conducted from May 2018 to April 2020. Patients with primary pterygium who attended eye clinic Hospital Universiti Sains Malaysia (HUSM) Kubang Kerian, Kelantan and fulfilled the inclusion and exclusion criteria were recruited as participants of this study. Convenient sampling method was applied for participants' recruitment where all patients will be given thorough explanation in regards to the study and subsequently divided into interventional and control group. Intervention group participants were given intralesional Ranibizumab (0.5mg/ 0.05mL) 2 weeks prior to pterygium excision surgery. Both groups of participants undergo pterygium excision with autologous conjunctival graft surgery thereafter. Excised pterygium tissues were sent to the laboratory for slide preparation and staining with specific reagents including Masson Trichrome for collagen fibers, anti CD34 antibody for microvascular density and anti-8 OHdG antibody for oxidative stress changes. Slides were then analysed by the pathologist and statistical analysis of the results were carried out with the Statistical Package for the Social Sciences (SPSS) Version 26.0. All participants had intralesional Ranibizumab injection and pterygium excision with autologous conjunctival graft surgery in May 2018. They were scheduled for follow-up visits for the next 24 months to observe for complications of intralesional Ranibizumab injection, pterygium excision and conjunctival autograft surgery and any signs of recurrence.

ELIGIBILITY:
Inclusion Criteria:

* primary nasal grade 2 to 3 pterygium based on the clinical stages outlined by Johnston et al (2004)
* who consented for pterygium excision and conjunctival autograft surgery

Exclusion Criteria:

* cornea pathology such as scarring, history of herpetic keratitis, eyelid abnormalities, previous ocular surgery, ocular trauma, and ocular or systemic inflammatory disease
* Pregnant women and lactating mothers

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Microvascular Density (MVD) using anti-CD34 antibody staining, classified based on the Weidner scoring system. | After pterygium excision surgery, tissues were sent to the histopathological laboratory where microvascular density was assessed within two weeks
  MVD is a reflection of angiogenesis (Norrby, 1998). The effects of anti-VEGF on MVD of the excised tissue were assessed using anti-CD34 antibody (50 µg at 1 mg/ml at dilution of 1:50-1:100, QBEnd/10, Mouse anti-Human, Dako, North America).

SECONDARY OUTCOMES:
Oxidative Stress using eight-hydroxyguanosine (8-OHdG) staining, based on the percentage of positively stained cells viewed under 400x high-power field magnification. | After pterygium excision surgery, tissues were sent to the histopathological laboratory where assessment for oxidative stress via 8-OHdG staining was performed within two weeks
  8-OHdG is an oxidative stress biomarker which has been observed to have a significant association with primary pterygium Ismaeel et al. (2010).

CONTACTS AND LOCATIONS:
Overall Officials: Jin Yi Yap, MMed, Principal Investigator — Universiti Sains Malaysia
Locations (1):
- Hospital Universiti Sains Malaysia, Kota Bharu, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ismaeel OM, Jaafar H, Ibrahim M. Detection of 8-hydroxydeoxyguanosine enzyme in recurrent pterygium raising a question on its role on recurrence. Int J Ophthalmol. 2010;3(3):245-8. doi: 10.3980/j.issn.2222-3959.2010.03.15. Epub 2010 Sep 18. PMID 22553564
- [Background] Johnston SC, Williams PB, Sheppard JDJr. A Comprehensive System for Pterygium Classification. Invest Ophthalmol Vis Sci. 2004; 45(13): 2940.
- [Background] Norrby K. Microvascular density in terms of number and length of microvessel segments per unit tissue volume in mammalian angiogenesis. Microvasc Res. 1998 Jan;55(1):43-53. doi: 10.1006/mvre.1997.2054. PMID 9473408
- [Background] Shibuya M. Vascular Endothelial Growth Factor (VEGF) and Its Receptor (VEGFR) Signaling in Angiogenesis: A Crucial Target for Anti- and Pro-Angiogenic Therapies. Genes Cancer. 2011 Dec;2(12):1097-105. doi: 10.1177/1947601911423031. PMID 22866201
- [Background] Karaman S, Leppanen VM, Alitalo K. Vascular endothelial growth factor signaling in development and disease. Development. 2018 Jul 20;145(14):dev151019. doi: 10.1242/dev.151019. PMID 30030240
- [Background] Cardenas-Cantu E, Zavala J, Valenzuela J, Valdez-Garcia JE. Molecular Basis of Pterygium Development. Semin Ophthalmol. 2016;31(6):567-83. doi: 10.3109/08820538.2014.971822. Epub 2014 Nov 21. PMID 25415268
- [Background] Rossino MG, Lulli M, Amato R, Cammalleri M, Monte MD, Casini G. Oxidative Stress Induces a VEGF Autocrine Loop in the Retina: Relevance for Diabetic Retinopathy. Cells. 2020 Jun 11;9(6):1452. doi: 10.3390/cells9061452. PMID 32545222